CLINICAL TRIAL: NCT03214107
Title: Comparison of Two Carbohydrate Intake Strategies to Improve Glucose Control During Exercise in Adolescents and Adults With Type 1 Diabetes
Brief Title: Carbohydrate-based Strategies to Prevent Exercise-induced Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Director of the Research Platform on Obesity, Metabolism and Diabetes, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SNACK-1
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Exercise; Hypoglycemia; Carbohydrates
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Exercise; Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full snack given before exercise (Active Comparator): A snack containing ~0.5g of carbohydrates per kilogram of body weight will be given 5 minutes before exercise
  Interventions: Other: Exercise; Other: Snack
- Distributed snack over exercise period (Active Comparator): A snack containing ~0.5g of carbohydrates per kilogram of body weight distributed this way will be given: ~40% given 5 minutes before exercise, ~30% after 20 minutes of exercise and the last ~30% after 40 minutes of exercise.
  Interventions: Other: Exercise; Other: Snack

INTERVENTIONS:
Other: Exercise — Participants will be admitted at IRCM at 14:00. At 15:30, participants will performed a 60-minute exercise on the ergocycle at 60% of VO2 peak (moderate intensity). During exercise, capillary glucose levels will be measured every 10 minutes. At 16:30, the exercise will be completed and capillary glucose levels will be monitored every 20 minutes for 1 hour. At 17:30, the participant will be discharged.
Other: Snack — Full snack or Distributed snack

SUMMARY:
To prevent hypoglycemia during prolonged exercise (>30 minutes), additional carbohydrate intake is frequently required. Carbohydrate intake required will vary with insulin regimens, timing and type of exercise as well as starting blood glucose level. In addition to the amount of carbohydrate ingested, the timing of carbohydrate intake could also have an impact on glucose control during exercise. Therefore, the objective of this study will be to compare the efficacy of two snacking strategies to maintain glucose levels in the target range during an exercise period in adolescents and adults with type 1 diabetes: 1) a snack containing ~0.5g of carbohydrates per kilogram of body weight - rounded to the nearest 5g - given 5 minutes before exercise; 2) a snack containing ~0.5g of carbohydrates per kilogram of body weight - rounded to the nearest 5g - distributed this way: ~40% given 5 minutes before exercise, ~30% after 20 minutes of exercise and the last ~30% after 40 minutes of exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 14 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. Last (less than 3 months) HbA1c ≤ 10%.
4. Patients using multiple daily injections with basal-bolus insulin regimen.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Abnormal blood panel and/or anemia.
4. Ongoing pregnancy.
5. Severe hypoglycemic episode within two weeks of screening.
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).
7. Treatment with CSII (Continuous Subcutaneous Insulin Infusion) "insulin pump therapy".

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Percentage of time of capillary glucose levels spent between 4-10 mmol/L | This outcome will be measured over 120 minutes
  This time frame corresponds to the exercise period and the 1 hour following it

SECONDARY OUTCOMES:
Percentage of time of sensor glucose levels spent between 4-10 mmol/L | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Percentage of time of glucose levels spent below 4 mmol/L | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Decrease in glucose levels | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
  Difference between glucose level at the start of the exercise and the lowest glucose level from the start of the exercise until 1) the end of the exercise and 2) 1 hour after the end of the exercise.
Increase in glucose level | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
  Difference between glucose level at the start of the exercise and the highest glucose level from the start of the exercise until 1) the end of the exercise and 2) 1 hour after the end of the exercise.
Number of participants with an exercise-induced hypoglycemia below 4 mmol/L | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Number of participants with an exercise-induced hypoglycemia below 3.5 mmol/L | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Number of participants requiring an oral treatment for hypoglycemia | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Total number of hypoglycemia episodes requiring treatment | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Percentage of time of glucose levels spent above 10 mmol/L | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Mean time (minutes) to the first hypoglycemic event | This outcome will be measured for the exercise period only (60 minutes)
Mean glucose levels | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Standard deviation of glucose levels | This outcome will be measured for the exercise period only (60 minutes) and for the exercise period and the hour following the exercise (120 minutes)
Percentage of time of glucose levels between 4 and 10 mmol/L | From the end of the exercise period to dinner time.
  Dinner time will be up to the patient.
Percentage of time of glucose levels between 4 and 10 mmol/L | From the end of the exercise period to midnight (7.5 hours)
Percentage of time of glucose levels between 4 and 10 mmol/L | From midnight to 6:00 next morning (6 hours)
Percentage of time of glucose levels between 4 and 10 mmol/L | From the end of the exercise period to 6:00 next morning (13.5 hours)
Percentage of time of glucose levels spent below 4 mmol/L | From the end of the exercise period to dinner time
  Dinner time will be up to the patient.
Percentage of time of glucose levels spent below 4 mmol/L | From the end of the exercise period to midnight (7.5 hours)
Percentage of time of glucose levels spent below 4 mmol/L | From midnight to 6:00 next morning (6 hours)
Percentage of time of glucose levels spent below 4 mmol/L | From the end of the exercise period to 6:00 next morning (13.5 hours)
Percentage of time of glucose levels spent above 10 mmol/L | From the end of the exercise period to dinner time
  Dinner time will be up to the patient
Percentage of time of glucose levels spent above 10 mmol/L | From the end of the exercise period to midnight (7.5 hours)
Percentage of time of glucose levels spent above 10 mmol/L | From midnight to 6:00 next morning (6 hours)
Percentage of time of glucose levels spent above 10 mmol/L | From the end of the exercise period to 6:00 next morning (13.5 hours)
Number of participants requiring treatment for hypoglycemia | From the end of the exercise period to dinner time
  Dinner time will be up to the patient
Number of participants requiring treatment for hypoglycemia | From the end of the exercise period to midnight (7.5 hours)
Number of participants requiring treatment for hypoglycemia | From midnight to 6:00 next morning (6 hours)
Number of participants requiring treatment for hypoglycemia | From the end of the exercise period to 6:00 next morning (13.5 hours)
Number of hypoglycemic episodes requiring treatment | From the end of the exercise period to dinner time
  Dinner time will be up to the patient
Number of hypoglycemic episodes requiring treatment | From the end of the exercise period to midnight (7.5 hours)
Number of hypoglycemic episodes requiring treatment | From midnight to 6:00 next morning (6 hours)
Number of hypoglycemic episodes requiring treatment | From the end of the exercise period to 6:00 next morning (13.5 hours)
Mean glucose levels | From the end of the exercise period to dinner time
  Dinner time will be up to the patient
Mean glucose levels | From the end of the exercise period to midnight (7.5 hours)
Mean glucose levels | From midnight to 6:00 next morning (6 hours)
Mean glucose levels | From the end of the exercise period to 6:00 next morning (13.5 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Goulet-Gelinas L, Saade MB, Suppere C, Fortin A, Messier V, Taleb N, Tagougui S, Shohoudi A, Legault L, Henderson M, Rabasa-Lhoret R. Comparison of two carbohydrate intake strategies to improve glucose control during exercise in adolescents and adults with type 1 diabetes. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1238-1246. doi: 10.1016/j.numecd.2020.12.011. Epub 2020 Dec 17. PMID 33632598